CLINICAL TRIAL: NCT05723419
Title: Perfusion Index Value in Predicting the Clinical Outcome of Axillary Block
Brief Title: Prediction of Clinical Outcome in Axillary Block
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 20201-025-04
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: axillary block using 5 ml local anesthetics — ultrasoud guided axillary block

SUMMARY:
The primary endpoint of this study was to identify that Perfusion index (PI) has any predictive value for the treatment outcome of cervical radiculopathy

DETAILED DESCRIPTION:
The interscalene brachial plexus block is an effective intervention for reducing postoperative pain but is related to side effects, Suprascapular nerve block and a block of the axillary nerve have been introduced as alternatives to the interscalene brachial plexus for the control of postoperative pain. Previous study demonstrated new method of axillary block using interfascial plane injection guided by ultrasoud. Axillary block has been used widely for the relief of postoperative arm pain.

Recent study deomonstrated good pain relief when ultrasound guided fascial plane injection was performed in patients with cervical radiuculopathy.

The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. Although the special probe for PI measurement is relatively more expensive compared with ordinary pulse oximetery probes, its benefit as a marker of peripheral perfusion and as an idex for sympathetic stimulation have increased its use progressively. PI has been used widely for the prediction of success of brachial plexus block or axillary block. Changes of PI ratio value showed an excellent predictive value for the success of block.

There have been no studies demonstrating any predictive value of PI in axillary block for the relief of cervical radiulopathy

ELIGIBILITY:
Inclusion Criteria:

* Cervical foraminal stenosis
* Cervical central stenosis
* Cervical disc herniation
* Cervical spondylolisthesis

Exclusion Criteria:

* Infection
* pregnancy
* allergy to local anesthetic agents
* previous cervical spine surgery

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who visit the pain clinic
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Perfusion index changes among 4 time periods | baseline, 10 minutes, 20 minutes, 30 minutes after axillary block
  Perfusion index changes among 4 time periods
Number of patients showing numerical rating scale reduction more than 50% | 1 month after axillary block
  Number of patients showing numerical rating scale reduction more than 50%
Number of patients showing numerical rating scale reduction less than 50% | 1 month after axillary block
  Number of patients showing numerical rating scale reduction less than 50%
Number of patients showing no reduction in numerical rating scale | 1 month after axillary block
  Number of patients showing no reduction in numerical rating scale
Neck disability index changes between 2 time periods | baseline, 1 month after axillary block
  Neck disability index changes between 2 time periods

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Hoon Park, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No